CLINICAL TRIAL: NCT03921814
Title: Clinical Investigation of Safety and Efficacy of a Philips Intense Pulsed Light Device for Hair Reduction (Sunstone 2019)
Brief Title: Sunstone IPL (Intense Pulsed Light) for Hair Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC-BEA-Sunstone-2018-10510
Record Dates: First submitted 2019-04-01; First posted 2019-04-19 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Hair Removal
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will be treated with the investigation device.
Masking Description: Periodic photographs are taken of the treatment areas. The photos are labeled with a randomized bar code label. Hair counters will review the photos and count the hairs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment with IPL device (Experimental): This study will be conducted in women, aged 18 to 65 years, with skin types I up to and including V, and measured melanin values of ≤ 553 Melanin index in each qualifying treatment area in face (upper lip), axilla, bikini line, and leg. Each of the 2cm x 4cm treatment area bilateral located in axilla, bikini line and leg should count a minimum of 24 hairs. In face (upper lip) on upper lip, a minimum of 10 hairs should be available in each of the 1cm x 2cm selected treatment area bilateral located. The procedure to define the treatment area is described in the Training Manual [5]. Skin type must be determined based on an evaluation by a dermatologist or designee at site according to the Fitzpatrick Skin Type Scale.
  Interventions: Device: Treatment with IPL device

INTERVENTIONS:
Device: Treatment with IPL device — Exposure of body parts to the IPL device

SUMMARY:
This is a prospective, multi-center, single-arm, single blinded study to evaluate the safety and efficacy of the Sunstone IPL (Intense Pulsed Light) device to remove hair.

DETAILED DESCRIPTION:
Prospective, multi-center, single-arm, single blinded (Philips hair counter) study in healthy women of skin types I up to and including V.

Safety and efficacy of hair removal with the Investigational Philips IPL-device will be investigated.

In-clinic, each study subject will undergo twelve IPL-treatments at four areas bilaterally (face, axilla, bikini line, and legs) with an investigational IPL device applied by a device operator.

Hair re-growth in four body areas, face, axillae, bikini line and leg will be evaluated separately.

After the 4 bi-weekly treatments, one follow-up visit will be organized. After the completion of full treatment cycle (12 treatments), subjects will be followed for 1 and 3 months (short-term follow-up) and for 6, 9 and 12 months (long-term follow up).

ELIGIBILITY:
Inclusion Criteria:

1. Be willing to provide informed consent
2. Have a minimum of 24 hairs in each of the 2x4cm2 treatment area in axilla, bikini line, and leg, by visual inspection
3. Have a minimum of 10 hairs in the 1x2cm2 treatment area in face (upper lip), by visual inspection
4. Have a Fitzpatrick Skin Type I to V, with a melanin index less or equal to 553, as measured by Mexameter MX 18 in the designated treatment areas on face, axilla, bikini, and legs
5. Have natural body hair color that is dark blonde to black in the designated treatment areas
6. Are female subjects 18-65 years of age
7. Be either post-menopausal or surgically sterilized, or using a medically acceptable form of birth control (e.g., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence, etc.).
8. Be willing to participate in all scheduled study visits
9. Be willing to refrain from deliberate exposure to strong sun, products or procedures that would cause the skin to become darker in the designated treatment areas during the treatment phase
10. Be willing to refrain from the use of hair growth inhibitors/accelerators during the course of the study
11. Be willing to refrain from waxing, depilating or epilating of the face (upper lip), axilla, bikini line, and leg during the course of the study
12. Be willing to refrain from using aspirin or NSAIDS (e.g. acetaminophen, ibuprofen, etc.) within 5 days prior to and 5 days after treatment(s)

Exclusion Criteria:

1. Have fewer than 8 qualifying treatment areas: 2 in face (upper lip), 2 in axilla, 2 on bikini line, 2 on leg)
2. Have a malignant or pre-malignant pigmented lesion in the area to be treated
3. Have scarring or infection of the area to be treated
4. Have a known history of photosensitivity or use of medication known to induce photosensitivity
5. Are currently pregnant or lactating or planning to become pregnant in the period of the study, per subject report
6. Are currently on a daily dose of aspirin or NSAIDS (e.g. acetaminophen, ibuprofen, etc.) or have taken aspirin and/or NSAID within 5 days prior to treatment that would reduce or increase the sensation of pain
7. Are not willing to abstain from the use of products or light exposure that would induce tanning in the treatment areas during the IPL treatment period (first 10 months)
8. Have a history of immunosuppressive disease (including HIV infection or AIDS)
9. Are on anticoagulative medication or have thromboembolic condition
10. Any form of isotretinoin (such as Accutane or Roaccutane etc.) in the last six months.
11. Have an active implantable device such as a pacemaker, neurostimulator or internal defibrillator
12. Have used waxing or other methods of root hair removal, or photo-epilation within 6 months prior to treatment
13. Have been exposed to strong sunlight or an artificial tanning machine within 4 weeks of enrolment
14. Have a tattoo(s), warts, moles, benign skin lesions, dark pigmented areas, permanent make-up etc. in the treatment areas.
15. Have eczema, psoriasis, lesions, open wounds or any skin affliction in the treatment areas
16. Have a history of keloid scar formation
17. Have a history of herpes outbreaks in the designated treatment areas
18. Have a history of photosensitive epilepsy
19. Have a condition related to hormonal changes like polycystic ovarian syndrome (PCOS) or taking drugs leading to hormonal changes resulting in excessive hair growth like hirsutism and idiopathic hirsutism
20. Have diabetes, or metabolic disease that affects hair growth
21. Taking immunosuppressive medication(s)
22. Have a disease related to photosensitivity, such as polymorphic light eruption (PMLE), solar urticaria, porphyria etc.
23. Have a history of skin cancer, including past basal cell carcinoma and/or squamous cell carcinoma in the designated treatment areas
24. Have a history of any radiation therapy in any of the designated treatment areas
25. Have a history of radiation therapy in non-treatment areas within 5 years
26. Have a history of chemotherapy
27. Have used hair growth inhibitors and/or accelerators within 6 months preceding enrolment
28. Have had laser or electrolysis treatment for the removal of hair in the treatment sites within the last year
29. Have natural body hair colors of white, grey, light to mid-blond, or red in the designated treatment areas
30. Have bleaching of the body hair in the designated treatment areas 6 months prior to study enrolment
31. Have shaved treatment areas within 7 days prior to study enrolment
32. Participating in other clinical studies prior to, or concurrently with this study, that could be deemed to interfere with full and complete participation in this study - as determined by the site Investigator.

    -

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety of the Sunstone IPL device on removal of unwanted hair on face, axillae, bikini area and legs over the course of the treatment (12 treatments) and follow up (12 months). | approximately 18 months
  The analysis of the Primary safety endpoint will be based on the safety population which include all the enrolled subjects with at least one treatment. The primary safety endpoints include the treatment-emerged, anticipated adverse events (e.g. pain/discomfort, anticipated skin reactions.), non-anticipated adverse events, serious adverse events and reasons for discontinuation. Pain/discomfort will be evaluated per treatment per body area using the 5-point pain score grade. The percentage of the top-two scores will be calculated. Skin reactions will be assessed per treatment and body area, and will be described for type, onset, duration and severity. Incidence of adverse events will be summarized by frequency, severity and by relationship to device. Safety data will be summarized with descriptive statistics by body area, time points and clinical sites and combined.
Evaluation of the efficacy of the Sunstone IPL device on short-term hair reduction on face, axillae, bikini area and legs, 1 month after the last treatment (12 treatments). | approximately 11 months
  The primary efficacy endpoint is the proportion of subjects with successful hair reduction at 1 month post-final treatment per body area. Successful hair reduction is defined as an average reduction in hair count at the given time point, that is greater than or equal to 30% relative to baseline hair count. Post-final treatment is defined as time point after the last of 12 treatments.
Evaluation of the efficacy of the Sunstone IPL device on short-term hair reduction on face, axillae, bikini area and legs, 3 months after the last treatment (12 treatments). | approximately 14 months
  The primary efficacy endpoint is the proportion of subjects with successful hair reduction at 3 months post-final treatment per body area. Successful hair reduction is defined as an average reduction in hair count at the given time point, that is greater than or equal to 30% relative to baseline hair count. Post-final treatment is defined as time point after the last of 12 treatments.

SECONDARY OUTCOMES:
4. Evaluation of the efficacy of the Sunstone IPL device on removal of unwanted hair on face, axillae, bikini area, and legs after the initial, intensive treatment phase at 8 weeks after baseline (2 weeks after the 4th treatment). | Approximately 2 months
  Proportion of subjects with successful hair reduction (greater than or equal to 30% relative to baseline) at 8 weeks post-baseline (2 weeks after the 4th treatment) per body area.
5. Evaluation of the efficacy of the Sunstone IPL device on removal of unwanted hair on face, axillae, bikini area, and legs after the initial, intensive treatment phase at 10 weeks after baseline (4 weeks after the 4th treatment). | Approximately 4.5 months
  Proportion of subjects with successful hair reduction (greater than or equal to 30% relative to baseline) at 10 weeks post-baseline (4 weeks after the 4th treatment) per body area.
6. Evaluation of the stable long-term hair reduction efficacy in face, axillae, bikini area and legs, 6, 9 and 12 months after completion of the 12 treatments with the Sunstone IPL device. | Approximately 22 months
  Proportion of subjects with successful hair reduction (greater than or equal to 30% relative to baseline) at 6, 9 and 12 months post-final treatment (12 treatments) per body area.
7. Assessment of the subjective satisfaction with the treatment results of the Sunstone IPL device s for removal of unwanted hair on face, axillae, bikini area, and legs. | Approximately 22 months
  Percent of top-two category answers of 5-point Likert satisfaction scale in assessment of subjective satisfaction with the treatment results in all body areas.
8. Assessment of the acceptance of the Philips investigational IPL devices for removal of unwanted hair in each body area. | Approximately 22 months
  Percent of top-two category answers in assessment of acceptance of hair reduction, skin smoothness, and comfort after treatment with Philips investigational IPL devices in all body areas.
Evaluate time course of hair reduction during first four treatments | Approximately 2 months
  Evaluate the time course of hair reduction to baseline achieved by the Philips investigational IPL device for each body area during the first four treatments, i.e. during the Intensive Treatment phase.

OTHER OUTCOMES:
Exploratory objective to assess subjective selection of setting compared to device setting | Approximately 18 months
  Exploratory objective:
  Assess the percentage of subjects who select a setting based on comfort, which is the same setting as indicated by the device.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Lotz, Study Director — Head of Global Clinical and Scientific Affairs
Locations (2):
- United States (2):
  - Sera Collection, Montebello, California
  - Sadick Research Group, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altshuler GB, Anderson RR, Manstein D, Zenzie HH, Smirnov MZ. Extended theory of selective photothermolysis. Lasers Surg Med. 2001;29(5):416-32. doi: 10.1002/lsm.1136. PMID 11891730
- [Background] Ravnbak MH. Objective determination of Fitzpatrick skin type. Dan Med Bull. 2010 Aug;57(8):B4153. PMID 20682135
- [Background] Shamsuddin K et. al, The reliability of Fitzpatrick Skin Type Chart Comparing to Mexameter (Mx 18) in measuring skin color among first trimester, Malaysian Journal of Public Health Medicine 2016, Vol. 16 (3): 59-65
- [Background] Town G, Ash C, Dierickx C, Fritz K, Bjerring P, Haedersdal M. Guidelines on the safety of light-based home-use hair removal devices from the European Society for Laser Dermatology. J Eur Acad Dermatol Venereol. 2012 Jul;26(7):799-811. doi: 10.1111/j.1468-3083.2011.04406.x. Epub 2012 Jan 3. PMID 22211702
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516